CLINICAL TRIAL: NCT07033286
Title: Early Esophagogastroduodenoscopy Performed Bedside Using Single-use Disposable Endoscope - A Prospective Non-randomized Controlled Single Centre Study
Brief Title: Early Esophagogastroduodenoscopy Performed Bedside Using Single-use Disposable Endoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Camilla Kjelkvist-Born, Principal Investigator, Zealand University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BedsideGAS_pilot
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Upper Gastrointestinal Disorder
Keywords: Gastroscopy; Upper endoscopy; Gastroscope; Esophagogastroduodenoscope; Single-use; Reusable; Bedside
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, quality assurance study. Non-randomized, controlled single center feasibility study. Comparing a period where subacute gastroscopies are performed in the endoscopy unit (reusable gastroscopes) with a period where they are performed bedside in the patients room (single-use gastroscopes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reusable gastroscope in the endoscopy unit (Active Comparator): In the first period the subacute gastroscopies will be performed with a reusable gastroscope in the endoscopy unit.
  Interventions: Device: Diagnostic gastroscopes, Olympus
- Single-use gastroscope bedside in the patient's room (Experimental): In the second period the subacute gastroscopies will be performed with a reusable gastroscope in bedside in the patients' rooms.
  Interventions: Device: Ambu aScope Gastro

INTERVENTIONS:
Device: Ambu aScope Gastro — CE-marked single-use gastroscopes from Ambu are used in the single-use group.
  Arms: Single-use gastroscope bedside in the patient's room
Device: Diagnostic gastroscopes, Olympus — Reusable gastroscopes from Olympus are used in the reusable group.
  Arms: Reusable gastroscope in the endoscopy unit

SUMMARY:
We aim to evaluate whether the use of single-use gastroscopes at the bedside can reduce the time from clinical indication to procedure compared to reusable gastroscopes used in the endoscopy unit for patients referred for subacute gastroscopy.

Participants in the first period will be scheduled for gastroscopy with a reusable gastroscope in the endoscopy unit, whereas participants during the second period will have a gastroscopy performed at the hospital department (bed-side) with a single-use gastroscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender, 18 years of age or older
* Diagnostic EGD without general anaesthesia

Exclusion Criteria:

* ASA-score of 4 or higher
* Unstable patient
* Suspicion of active bleeding
* Anticoagulants not withheld due to regional guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
Time from the indication/decision for early endoscopy to procedure | From indication to procedure, up to two weeks
Endoscopists' rating of the gastroscope | Immediately after procedure
  The endoscopists' rating of the gastroscope

SECONDARY OUTCOMES:
Time from admission to procedure | From admission to procedure, up to 3 months
Time from procedure to discharge | From procedure to discharge, up to 3 months
Duration of the procedure | During the procedure
Did the patient need sedation or local anaesthetic throat spray? | During the procedure
  Frequency of use of sedation and/or local anaesthetic throat spray in each group.
Technical success | From admission to discharge, up to 3 months
  Technical success is defined as the ability to complete the procedure adequately based on the indication and guidelines.
Complications to gastroscopy | 24 and 72 hour follow-up after procedure
Need for converting to general anaesthesia or reusable gastroscope | During admission, up to 3 months
  Did the patient need a new gastroscopy during admission? If so, what is the reason for that, according to the patient's medical record?
Findings during the procedure | During the procedure
  The frequency of various findings observed during the procedure in each group (e.g., gastric ulcer, varices, stenosis), based on the procedure documentation in the patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Bulut, Study Director — Surgical department of Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slivka A, Ross AS, Sejpal DV, Petersen BT, Bruno MJ, Pleskow DK, Muthusamy VR, Chennat JS, Krishnamoorthi R, Lee C, Martin JA, Poley JW, Cohen JM, Thaker AM, Peetermans JA, Rousseau MJ, Tirrell GP, Kozarek RA; EXALT Single-use Duodenoscope Study Group. Single-use duodenoscope for ERCP performed by endoscopists with a range of experience in procedures of variable complexity. Gastrointest Endosc. 2021 Dec;94(6):1046-1055. doi: 10.1016/j.gie.2021.06.017. Epub 2021 Jun 26. PMID 34186052
- [Background] Muthusamy VR, Bruno MJ, Kozarek RA, Petersen BT, Pleskow DK, Sejpal DV, Slivka A, Peetermans JA, Rousseau MJ, Tirrell GP, Ross AS. Clinical Evaluation of a Single-Use Duodenoscope for Endoscopic Retrograde Cholangiopancreatography. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2108-2117.e3. doi: 10.1016/j.cgh.2019.10.052. Epub 2019 Nov 6. PMID 31706060
- [Background] Bai Z, Wang R, Cheng G, Ma D, Ibrahim M, Chawla S, Qi X. Outcomes of early versus delayed endoscopy in cirrhotic patients with acute variceal bleeding: a systematic review with meta-analysis. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e868-e876. doi: 10.1097/MEG.0000000000002282. PMID 35048654
- [Background] Gralnek IM, Camus Duboc M, Garcia-Pagan JC, Fuccio L, Karstensen JG, Hucl T, Jovanovic I, Awadie H, Hernandez-Gea V, Tantau M, Ebigbo A, Ibrahim M, Vlachogiannakos J, Burgmans MC, Rosasco R, Triantafyllou K. Endoscopic diagnosis and management of esophagogastric variceal hemorrhage: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2022 Nov;54(11):1094-1120. doi: 10.1055/a-1939-4887. Epub 2022 Sep 29. PMID 36174643
- [Background] Jeong N, Kim KS, Jung YS, Kim T, Shin SM. Delayed endoscopy is associated with increased mortality in upper gastrointestinal hemorrhage. Am J Emerg Med. 2019 Feb;37(2):277-280. doi: 10.1016/j.ajem.2018.05.049. Epub 2018 May 24. PMID 29848459
- [Background] Siau K, Hodson J, Ingram R, Baxter A, Widlak MM, Sharratt C, Baker GM, Troth T, Hicken B, Tahir F, Magrabi M, Yousaf N, Grant C, Poon D, Khalil H, Lee HL, White JR, Tan H, Samani S, Hooper P, Ahmed S, Amin M, Mahgoub S, Asghar K, Leet F, Harborne MJ, Polewiczowska B, Khan S, Anjum MR, McFarlane M, Mozdiak E, O'Flynn LD, Blee IC, Molyneux RM, Kurian A, Abbas SN, Abbasi A, Karim A, Yasin A, Khattak F, White J, Ahmed R, Morgan JA, Alleyne L, Alam MA, Palaniyappan N, Rodger VJ, Sawhney P, Aslam N, Okeke T, Lawson A, Cheung D, Reid JP, Awasthi A, Anderson MR, Timothy JR, Pattni S, Ahmad S, Townson G, Shearman J, Giljaca V, Brookes MJ, Disney BR, Guha N, Thomas T, Norman A, Wurm P, Shah A, Fisher NC, Ishaq S, Major G. Time to endoscopy for acute upper gastrointestinal bleeding: Results from a prospective multicentre trainee-led audit. United European Gastroenterol J. 2019 Mar;7(2):199-209. doi: 10.1177/2050640618811491. Epub 2018 Oct 28. PMID 31080604
- [Background] Garg SK, Anugwom C, Campbell J, Wadhwa V, Gupta N, Lopez R, Shergill S, Sanaka MR. Early esophagogastroduodenoscopy is associated with better Outcomes in upper gastrointestinal bleeding: a nationwide study. Endosc Int Open. 2017 May;5(5):E376-E386. doi: 10.1055/s-0042-121665. PMID 28512647
- [Background] Gralnek IM, Stanley AJ, Morris AJ, Camus M, Lau J, Lanas A, Laursen SB, Radaelli F, Papanikolaou IS, Curdia Goncalves T, Dinis-Ribeiro M, Awadie H, Braun G, de Groot N, Udd M, Sanchez-Yague A, Neeman Z, van Hooft JE. Endoscopic diagnosis and management of nonvariceal upper gastrointestinal hemorrhage (NVUGIH): European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2021. Endoscopy. 2021 Mar;53(3):300-332. doi: 10.1055/a-1369-5274. Epub 2021 Feb 10. PMID 33567467